CLINICAL TRIAL: NCT00020930
Title: Phase II Study of an Anti-Epidermal Growth Factor Receptor (EGFR) Antibody, Cetuximab, in Patients With Irinotecan-Refractory, Stage IV Colorectal Carcinoma
Brief Title: Cetuximab in Treating Patients With Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068731; MSKCC-01034; IMCL-CP02-0141; NCI-G01-1970
Record Dates: First submitted 2001-07-11; First posted 2004-03-17 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab

INTERVENTIONS:
Biological: cetuximab

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of cetuximab in treating patients who have stage IV colorectal cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with irinotecan-refractory, stage IV colorectal cancer when treated with cetuximab. II. Determine the safety and toxic effects of this drug in these patients. III. Determine the time to progression of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive cetuximab IV over 1-2 hours weekly for 6 weeks. Treatment repeats in the absence of disease progression or unacceptable toxicity. Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent stage IV colorectal cancer Any T, any N, M1 Documented progressive disease within 6 months of completing an irinotecan- containing regimen Bidimensionally measurable metastatic disease Meningeal or CNS involvement allowed Immunohistochemical evidence of EGFR expression (at least 1+)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST no greater than 5 times ULN Alkaline phosphatase no greater than 5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No history of uncontrolled angina, arrhythmias, or congestive heart failure Other: No other malignancy within the past 3 years except basal cell skin cancer or pre-invasive carcinoma of the cervix No uncontrolled seizure disorder No neuropathy greater than grade 2 or other neurologic disease No medical or psychiatric condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior murine monoclonal antibody therapy or cetuximab Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy No other chemotherapy since completing irinotecan-containing regimen No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 30 days since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 21 days since prior surgery, except diagnostic biopsy, and recovered Other: At least 30 days since prior investigational agents and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States